CLINICAL TRIAL: NCT01707927
Title: Comparison of Two Biological Aortic Valves. Mosaic Ultra and Trifecta.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Bjørn Braathen, MD. Ph.D, Oslo University Hospital
Other Study IDs: 2011/2596/REK
Record Dates: First submitted 2012-09-12; First posted 2012-10-16 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Aortic Valve Stenosis
Keywords: EOA
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Trifecta: Degenerated aortic valve with indication for aortic valve replacement
- mosaic Ultra: Need a aortic valve replacement

SUMMARY:
Comparing two biological valves in a prospective randomized study. Mosaic Ultra and Trifecta. The investigators are looking at EOA and the Pressure Gradients over the valve by patients with the same annulus measured by a hegar dilatator.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve disease

Exclusion Criteria:

1. Pregnant
2. Breast feeding
3. Aortic valve bigger than 23 mm
4. Endocarditis
5. EF < 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated elektively for aortic valve disease with the need of a biological valve
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pressure gradients | 240 days
  Investigators want too look at the effient opening area and pressure gradients of the two valves we are implanting on patients with the same size of the annulus.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Braathen, MD Ph.D, Principal Investigator — OUS Thoraxkirurgisk avdeling Ullevål; Theis Tønnessen, MD Ph.D, Study Director — OUS thoraxkirurgisk avdeling Ullevål
Locations (1):
- Oslo university hospital, Thoracic departement, Oslo, Norway